CLINICAL TRIAL: NCT05487131
Title: Neuromodulation and Fatigue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: 14921
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Healthy Aging; Fatigue
Keywords: Transcutaneous spinal direct current stimulation; TsDCS; Fatigability
MeSH Terms: conditions — Fatigue | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Men (Experimental): Individuals will participate in 1 familiarization and 3 test sessions
  Interventions: Behavioral: electrical stimulation
- Women (Experimental): Individuals will participate in 1 familiarization and 3 test sessions
  Interventions: Behavioral: electrical stimulation

INTERVENTIONS:
Behavioral: electrical stimulation — different types of weak electrical stimulation will be used

SUMMARY:
In this project, we aim to determine any potential effects of a weak electrical current applied to the neck or thoracic area on functional capacity and muscle activation. Healthy individuals will participate in one familiarization followed by three experimental sessions. Fatigability and motor function will be assessed in each test session.

ELIGIBILITY:
Inclusion Criteria:

Healthy individuals between 18 and 50 years old

Exclusion Criteria:

Metal implants or joint replacement. Presence of neuromuscular disease. Skin hypersensitivity.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-03 (Actual); Primary Completion 2025-09-29 (Estimated); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Force | Each session will take approximately 2 hours (total of 4 test sessions)
  Change in force will be evaluated with a device during each test session
Perception of effort | Each session will take approximately 2 hours (total of 4 test sessions)
  Change in perceived effort will be evaluated with visual analogue scales
Muscle activation | Each session will take approximately 2 hours (total of 4 test sessions)
  Electromyography will be used to quantify muscle activation

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Pereira, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma, Norman, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No